CLINICAL TRIAL: NCT03457103
Title: Capnometry-Assisted Breathing Training for COPD
Acronym: CATCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-01672
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CATCH Group (Experimental): A portable capnometer (CapnoTrainer, Better Physiology, Cheyenne, WY) will be used in-session to provide continuous visual feedback of RR, ETCO2, rhythm, and depth of breathing, and ratio of inspirations to expiration. CATCH will be once weekly for 6 weeks, for a total of 6 sessions; each session will be approximately 60 minutes duration. The principal investigator will implement the CATCH intervention
  Interventions: Device: Capnometry-Assisted Training for COPD to Slow the Breath (CATCH); Device: Pulmonary Rehabilitation (PR)
- Control Group (Active Comparator): Pulmonary Rehabilitation (PR). Patients in both treatment groups will participate in a 10-week (16 - 20 sessions) comprehensive PR program.
  Interventions: Device: Pulmonary Rehabilitation (PR)

INTERVENTIONS:
Device: Capnometry-Assisted Training for COPD to Slow the Breath (CATCH) — Tailored intervention emphasizing slow, quiet, regular nasal breathing pattern.
  Arms: CATCH Group
Device: Pulmonary Rehabilitation (PR) — Patients in both treatment groups will participate in a 10 week (16-20 sessions) comprehensive PR program. The control group will receive the 10-Week PR program with traditional breathing training sessions (without biofeedback). The program comprises 2 or 3 exercise training sessions per week by physical therapists (each 1 hour duration).

SUMMARY:
Capnometry-Assisted Breathing Training for COPD (CATCH) is a behavioral intervention that aims to promote optimal, self-regulated, mindful breathing. A portable capnometer is used in-session to provide continuous visual feedback of Respiratory Rate (RR), End-Tidal Carbon Dioxide Tension (ETCO2), and breathing pattern. The tailored CATCH intervention will emphasize a slow, quiet, regular, nasal breathing pattern, as well as pursed lips breathing (PLB). CATCH is once weekly for 6 weeks, for a total of 6 sessions; each session is approximately 60 minutes long. The principal investigator will implement the CATCH intervention. The principal investigator will implement the CATCH intervention. Patients will use the Address Stress app on a smart phone or computer tablet as part of their home breathing exercises.

ELIGIBILITY:
Inclusion Criteria:

* over 40 years of age
* has COPD documented in their electronic medical record, as defined by FEV1/FVC of < 0.70 on pulmonary function testing (spirometry), or as shown on a chest CT
* Can maintain oxygen saturation (SaO2) ≥ 90% on room air at rest
* Is medically cleared to participate in NYULMC's outpatient pulmonary rehabilitation program
* English speaking. Pregnant patients will not be enrolled in the study

Exclusion Criteria:

* Requires 24-hour supplemental oxygen
* Has cognitive impairment as measured by ≤23/30 on the Mini Mental State Examination (MMSE)
* Is actively being treated for lung cancer (E.g. with chemotherapy or upcoming surgery)
* Has morbid obesity (BMI > 40)
* Is currently smoking
* Has unstable cardiac disease defined by a history of a myocardial infarction in the past 3 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Norweg, MD, Study Director — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Norweg AM, Wu Y, Troxel A, Whiteson JH, Collins E, Haas F, Skamai A, Goldring R, Jean-Louis G, Reibman J, Ehrlich-Jones L, Simon N. Mind-Body Intervention for Dysfunctional Breathing in Chronic Obstructive Pulmonary Disease: Feasibility Study and Lessons Learned. J Integr Complement Med. 2023 Mar;29(3):156-168. doi: 10.1089/jicm.2022.0552. Epub 2023 Feb 17. PMID 36800224

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CATCH Group | Control Group
Started | 22 | 9
Completed | 14 | 3
Not Completed | 8 | 6
Not completed — illness/hospitalization | 4 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — financial/ insurance issues | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CATCH Group | Control Group | Total
Number analyzed (Participants) | 22 | 9 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (10.45) | 71.4 (7.62) | 72.1 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 18
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 19 | 9 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 17 | 7 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adherence to Home Breathing Exercises
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | CATCH Group | Control Group
Number analyzed (Participants) | 14 | 5
Participants | 10 | 5

2. Secondary Outcome: Difference in Mean 6MWT Distance Between Pre and Post Intervention
Description: The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Time Frame: Week 0 and Week 10
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | CATCH Group | Control Group
Number analyzed (Participants) | 12 | 4
meters | 39.37 [14.13 to 64.61] | 24.99 [-32.53 to 82.52]

3. Secondary Outcome: Difference in Mean Dyspnea Management Questionnaire Computer Adaptive Test (DMQ-CAT) Anxiety Score Between Pre and Post Intervention
Description: The DMQ-CAT Dyspnea Anxiety is a 14 item scale; each item is scored off a 7 point likert scale for a total range of 0 to 98 where higher scores correlate with higher anxiety
Time Frame: 2 weeks pre intervention and 4 weeks post intervention
Population: -3.16 (-8.89, 2.57)
Measure: Mean (95% Confidence Interval); unit: score on DMQ-CAT (Anxiety)
Arm/Group | CATCH Group | Control Group
Number analyzed (Participants) | 13 | 3
score on DMQ-CAT (Anxiety) | 2.43 [.09 to 4.77] | -3.16 [-8.89 to 2.57]

4. Secondary Outcome: Mean Difference in Heart Rate Maximum Between Pre and Post Intervention
Time Frame: 0 weeks and 10 weeks
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | CATCH Group | Control Group
Number analyzed (Participants) | 10 | 2
beats per minute | 6.2 [-1.32 to 13.72] | 3 [-35.12 to 41.12]

5. Secondary Outcome: Difference in Mean PROMIS Fatigue Score Between Pre and Post Intervention
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue 7a questionnaire. Raw scores range from 7-35, with higher scores indicating higher levels of fatigue.
Time Frame: 0 weeks and 10 weeks
Measure: Mean (95% Confidence Interval); unit: score on PROMIS questionnaire
Arm/Group | CATCH Group | Control Group
Number analyzed (Participants) | 13 | 3
score on PROMIS questionnaire | -4.18 [-8.16 to -0.21] | 5.2 [-21.39 to 31.79]

6. Secondary Outcome: Mean Difference in Resting Respiratory Rate Between Pre and Post Intervention
Time Frame: 0 weeks and 10 weeks
Measure: Mean (95% Confidence Interval); unit: Breaths per minute
Arm/Group | CATCH Group | Control Group
Number analyzed (Participants) | 10 | 2
Breaths per minute | -2.75 [-7.56 to 2.05] | -4.2 [-26.26 to 17.87]

7. Secondary Outcome: Difference in Mean Score on St George's Respiratory Questionnaire (SGRQ) Between Pre and Post Intervention
Description: Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Time Frame: Week 0 and Week 10
Measure: Mean (95% Confidence Interval); unit: score on SGRQ questionnaire
Arm/Group | CATCH Group | Control Group
Number analyzed (Participants) | 12 | 3
score on SGRQ questionnaire | -11.76 [-19.68 to -3.83] | -9.96 [-38.07 to 18.14]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | CATCH Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/9
Other Adverse Events (participants affected / at risk) | 0/22 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT03457103/Prot_SAP_000.pdf